CLINICAL TRIAL: NCT01669226
Title: A Phase II,Randomized Study of an Addition Intraperitoneal Cisplatin and Etoposide to Standard First-line Therapy in Stage IIIC and Stage IV Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancer (EOC, FTC, PPC)
Brief Title: First-line Intraperitoneal Cisplatin and Etoposide Chemotherapy for Ovarian Cancer
Acronym: AICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Fudan University (Other); Shanghai Jiao Tong University School of Medicine (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01-2009-03; SGOG OV1 (Other: SGOG)
Record Dates: First submitted 2012-08-08; First posted 2012-08-20 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Bulky Stage IIIC and IV Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian Cancer; intraperitoneal chemotherapy
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Platinum; Etoposide; taxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen B, PEip and TCiv therapy (Experimental): Weekly IP cisplatin plus etoposide followed by IV paclitaxel plus carboplatin or docetaxel plus carboplatin
  Interventions: Drug: PEip (weekly) and TCiv
- Regimen A: Standard TCiv therapy (Active Comparator): IV paclitaxel plus carboplatin or docetaxel plus carboplatin
  Interventions: Drug: TCiv

INTERVENTIONS:
Drug: PEip (weekly) and TCiv — IP: cisplatin 50mg/m2 and etoposide 100mg/m2, weekly, 4 times; 14 days later IV: paclitaxel 175mg/m2 plus carboplatin AUC 5 or docetaxel 60-75mg/m2 plus carboplatin AUC 5
  Other Names: platinum; VP 16; taxane
  Arms: Regimen B, PEip and TCiv therapy
Drug: TCiv — IV: paclitaxel 175mg/m2 plus carboplatin AUC 5 or docetaxel 60-75mg/m2 plus carboplatin AUC 5
  Other Names: taxane; platinum
  Arms: Regimen A: Standard TCiv therapy

SUMMARY:
The purpose of this study is to evaluate the role of an additional intraperitoneal chemotherapy with cisplatin and etoposide in bulky advanced epithelial ovarian cancer.

DETAILED DESCRIPTION:
This exploratory trial is to compare the efficacy of sequential chemotherapy, intraperitoneal chemotherapy followed by intravenous chemotherapy, versus intravenous chemotherapy alone in the first-line therapy for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years to ≤ 75 years.
* Epithelial ovarian cancer with pathology confirmed stage IIIc or IV, expect for lymph node metastasis alone
* Optimal cytoreductive surgery, including hysterectomy, bilateral salpinges-oophorectomy, omentectomy, and resection of all metastatic lesions, with a residual disease no more than 1cm
* Available to receive intraperitoneal chemotherapy 5-10 days postoperative, or no more than postoperative 14 days for those with bowel resection.
* ECOG performance 0-2.
* No more than 3 cycles of chemotherapy prior to surgery.
* Laboratory testing within 7 days of registration: hematopoietic: absolute neutrophil count greater than 1,500/mm3; Platelet count greater than 100,000/mm3. Hepatic: bilirubin less than 1.25 times upper limit of normal (ULN); Bilirubin < 2.0, SGPT less than 2 times ULN. Renal: creatinine less than 1.6 mg/dL, OR creatinine clearance greater than 40 mL/min.
* Comply with intraperitoneal chemotherapy and follow-up.
* Written informed consent.

Exclusion Criteria:

* Low-malignant potential ovarian tumor.
* Laboratory testing insufficiency. Hemoglobin < 10 g/dL. Renal insufficiency with serum creatinine > 1.6.
* Bone marrow dysfunction: absolute neutrophil count less than 1,500/mm3; Platelet count less than 80,000/mm3.
* Active infection.
* Clinically significant gastrointestinal abnormalities.
* Active coronary artery disease, cerebrovascular disease, restrictive or obstructive pulmonary disease, or congestive heart failure.
* Other condition that could interfere with provision of informed consent, compliance to study procedures, or follow-up.
* Prior invasive malignancies within the last 5 years showing activity of disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-04; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
12-month disease non-progression rate | 12 months

SECONDARY OUTCOMES:
Progression-free survival | up to 120 months
Completion rate of intraperitoneal chemotherapy. | up to 6 months
Quality of life assessments | baseline; 4th week of intraperitoneal,chemotherapy, 6th cycle of intravenous chemotherpy, 3, 6, and 12 months after first-line chemotherapy.
Overall Survival | up to 120 months
adverse effects | Participants will be followed for the duration of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rongyu Zang, MD,PhD, Principal Investigator — Shanghai Gynecologic Oncology Group
Locations (7):
- China (7):
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Wuxi Cancer Hospital, Wuxi, Jiangsu
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Ren Ji Hospital Affiliated to Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Frist Maternity and Infant Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Fudan University Cancer Hospital, Shanghai

REFERENCES:
- [Derived] Shi T, Jiang R, Pu H, Yang H, Tu D, Dai Z, Cai Y, Zhang Y, Cheng X, Jia H, Tu R, Wang H, Tang J, Luan Y, Cai S, Zang R; SGOG-OV/AICE Investigators. Survival benefits of dose-dense early postoperative intraperitoneal chemotherapy in front-line therapy for advanced ovarian cancer: a randomised controlled study. Br J Cancer. 2019 Aug;121(5):425-428. doi: 10.1038/s41416-019-0543-1. Epub 2019 Aug 6. PMID 31383985
- See also: Shanghai Gynecologic Oncology Group — http://www.ShanghaiGOG.org